CLINICAL TRIAL: NCT04890990
Title: Reducing Depression-related Stigma and Increasing-treatment Seeking Among Black Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000028980
Record Dates: First submitted 2021-05-12; First posted 2021-05-18 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Depression; Racism
MeSH Terms: conditions — Depression; Racism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Black girl, control (BC) (Active Comparator): ~120-second video of a Black adolescent girl, without depression
  Interventions: Behavioral: Short videos
- Black girl, depressed (BD) (Active Comparator): ~120-second video of a Black adolescent girl, depressed
  Interventions: Behavioral: Short videos
- Black girl, depressed, adjusted (BDa) (Active Comparator): ~120-second video of a Black adolescent girl, depressed - adjusted for the specifics of being a Black girl (as informed by a focus group of Black girls and women)
  Interventions: Behavioral: Short videos

INTERVENTIONS:
Behavioral: Short videos — Intervention videos will each be of 90-second duration and feature two underage professionals (ages 16) acting as a simulated patient. All videos will focus on an empowered presenter with depression sharing her personal story regarding depression and describe how social supports from family, friends, and community, as well as professional help assisted her in overcoming symptoms of the illness. The actors will include a Black girl and a white girl.

SUMMARY:
The purposes of this study are to:

1. test among adolescent the utility of brief video-based interventions to reduce stigma-related attitudes and increase help-seeking intentions toward depression;
2. examine the role of race (Black vs other) as an independent factor in the primary outcome.

DETAILED DESCRIPTION:
Intervention videos will each be of ~120-second duration and feature an underage female professional (age 16) acting as a simulated patient. All three videos will focus on her as an empowered presenter with depression sharing her personal story regarding depression and describe how social supports from family, friends, and community, as well as professional help assisted her in overcoming symptoms of the illness.

Assessments will occur at baseline and post-intervention, and will include:

1. Demographics (baseline only);
2. Primary outcome: Depression-related stigma(Depression Stigma Scale [DSS]) summary score.
3. Secondary outcomes: a. DSS individual items; b. Help-seeking (General Help-Seeking Questionnaire [GHSQ]) summary score and individual items; and bc Racial attitudes: feelings thermometers.

The investigators intend to randomly assign ~1,000 individuals aged 14-18 as follows:

Subjects oversampled for Black participants (50% Black; 50% other);

Randomized, in equal proportions, and stratified by race, to view one of three ~120-second videos of a girl with:

1. No depression control (Black; BC);
2. Depression (Black, following same script as in our earlier study (Amsalem and Martin, 2021), DB); and
3. Depression adjusted (Black, with script adjusted based on input from focus group of Black girls and women; DBa).

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Living in the US
* Ages 14 - 18

Exclusion Criteria:

* None

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1291 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-08-07 (Actual); Study Completion 2021-08-07 (Actual)

PRIMARY OUTCOMES:
Change in Depression-related stigma (Depression Stigma Scale [DSS]; Personal component only): TOTAL SCORE | Before / after viewing videos (within 10 minutes)
  The DSS (Christensen, Jorm, Evans, & Groves, 2004) is a self-report instrument composed of two 9-item subscales. The first subscale measures the participants' own/ personal attitudes, and the second measures participants' beliefs about the attitudes of others ('Depression is sign of weakness' vs. 'Most people believe that depression is a sign of weakness'). We will use the Personal subscale (DSS-Personal) in this study. The DSS has a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). The total score comprises the sum of its item scores, and a higher score indicates more stigma (worse outcome). The DSS-Personal subscale has shown adequate psychometric properties: 0.71 test-retest reliability, 0.76 internal consistency (Griffiths et al., 2004). In our earlier study (Amsalem and Martin, 2021), Cronbach's a was .83.

SECONDARY OUTCOMES:
Change in Help-seeking (General Help-Seeking Questionnaire [GHSQ]; Emotional and Suicide components): MEAN SCORE | Before / after viewing videos (within 10 minutes)
  The General Help-Seeking Questionnaire (GHSQ) (Wilson, Deane, Marshall, & Dalley, 2008) was developed to measure help-seeking intentions from different sources (friend, parent, mental health professional, and others) and is divided into personal-emotional problems and suicidal thoughts (Ibrahim et al., 2019). The instrument consists of 10 items for each part, measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). One question is stated as 'I would not seek help from anyone' and is reverse-scored. Higher scores on this scale indicate more help seeking (better outcome). The GHSQ has shown good psychometric properties: Cronbach's alpha = .70 and test-retest of .86 for personal-emotional problems, and Cronbach's alpha = .83 and test-retest of .88 for suicidal thoughts.
Change in Racial attitudes: feelings thermometer | Before / after viewing videos (within 10 minutes)
  We will use a feelings thermometer, modeled after Norton and Herek, 2013:
  "Using a scale from zero to 100, please tell us your personal feelings toward each of the following groups of friends, teachers, or colleagues. As you do this task, think of an imaginary thermometer. The warmer or more favorable you feel toward the group, the higher the number you should give it. The colder or less favorable you feel, the lower the number. If you feel neither warm nor cold toward the group, rate it 50." To familiarize respondents with the response format, they will be first presented with thermometers for "Men in general" and "Women in general," with each respondent rating her or his own sex first. Next, they rate racially different groups (white women, white men, Black women, Black men) with the order of presentation randomized. Higher ratings (maximum 100) indicate warmer, more favorable feelings toward the target whereas lower ratings (minimum 0) indicate colder, more negative feelings.
Change in DSS Item 1 | Before / after viewing videos (within 10 minutes)
  People with depression could snap out of it if they wanted
  Scored on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). A higher score indicates more stigma (worse outcome).
Change in DSS Item 2 | Before / after viewing videos (within 10 minutes)
  Depression is a sign of personal weakness
  Scored on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). A higher score indicates more stigma (worse outcome).
Change in DSS Item 3 | Before / after viewing videos (within 10 minutes)
  Depression is not a real medical illness
  Scored on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). A higher score indicates more stigma (worse outcome).
Change in DSS Item 4 | Before / after viewing videos (within 10 minutes)
  People with depression are dangerous
  Scored on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). A higher score indicates more stigma (worse outcome).
Change in DSS Item 5 | Before / after viewing videos (within 10 minutes)
  It is best to avoid people with depression, so you don't become depressed yourself
  Scored on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). A higher score indicates more stigma (worse outcome).
Change in DSS Item 6 | Before / after viewing videos (within 10 minutes)
  People with depression are unpredictable
  Scored on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). A higher score indicates more stigma (worse outcome).
Change in DSS Item 7 | Before / after viewing videos (within 10 minutes)
  If I had depression, I would not tell anyone
  Scored on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). A higher score indicates more stigma (worse outcome).
Change in DSS Item 8 | Before / after viewing videos (within 10 minutes)
  I would not employ someone if I knew they had been depressed
  Scored on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). A higher score indicates more stigma (worse outcome).
Change in DSS Item 9 | Before / after viewing videos (within 10 minutes)
  I would not vote for a politician if I knew they had been depressed
  Scored on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). A higher score indicates more stigma (worse outcome).
Change in GHSQ Emotional Item 1 | Before / after viewing videos (within 10 minutes)
  Intimate partner (e.g., girlfriend, boyfriend)
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Emotional Item 2 | Before / after viewing videos (within 10 minutes)
  Friend (not related to you)
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Emotional Item 3 | Before / after viewing videos (within 10 minutes)
  Parent
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Emotional Item 4 | Before / after viewing videos (within 10 minutes)
  Other relative/family member
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Emotional Item 5 | Before / after viewing videos (within 10 minutes)
  Mental health professional (e.g., psychologist, social worker, counselor)
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Emotional Item 6 | Before / after viewing videos (within 10 minutes)
  Phone helpline (e.g., lifeline)
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Emotional Item 7 | Before / after viewing videos (within 10 minutes)
  Doctor/GP
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Emotional Item 8 | Before / after viewing videos (within 10 minutes)
  Minister or religious leader (e.g., Priest, Rabbi, Chaplain)
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Emotional Item 9 | Before / after viewing videos (within 10 minutes)
  I would not seek help from anyone
  **REVERSE SCORED ITEM** Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). LOWER scores on this item indicate more help seeking (better outcome).
Change in GHSQ Emotional Item 10 | Before / after viewing videos (within 10 minutes)
  I would seek help from another not listed above
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Suicide Item 1 | Before / after viewing videos (within 10 minutes)
  Intimate partner (e.g., girlfriend, boyfriend)
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Suicide Item 2 | Before / after viewing videos (within 10 minutes)
  Friend (not related to you)
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Suicide Item 3 | Before / after viewing videos (within 10 minutes)
  Parent
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Suicide Item 4 | Before / after viewing videos (within 10 minutes)
  Other relative/family member
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Suicide Item 5 | Before / after viewing videos (within 10 minutes)
  Mental health professional (e.g., psychologist, social worker, counselor)
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Suicide Item 6 | Before / after viewing videos (within 10 minutes)
  Phone helpline (e.g., lifeline)
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Suicide Item 7 | Before / after viewing videos (within 10 minutes)
  Doctor/GP
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Suicide Item 8 | Before / after viewing videos (within 10 minutes)
  Minister or religious leader (e.g., Priest, Rabbi, Chaplain)
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).
Change in GHSQ Suicide Item 9 | Before / after viewing videos (within 10 minutes)
  I would not seek help from anyone
  **REVERSE SCORED ITEM** Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). LOWER scores on this item indicate more help seeking (better outcome).
Change in GHSQ Suicide Item 10 | Before / after viewing videos (within 10 minutes)
  I would seek help from another not listed above
  Measured with a 7-point Likert scale ranging from 1 (extremely unlikely) to 7 (extremely likely). Higher scores on this item indicate more help seeking (better outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Griffiths KM, Christensen H, Jorm AF, Evans K, Groves C. Effect of web-based depression literacy and cognitive-behavioural therapy interventions on stigmatising attitudes to depression: randomised controlled trial. Br J Psychiatry. 2004 Oct;185:342-9. doi: 10.1192/bjp.185.4.342. PMID 15458995
- [Background] Wilson CJ, Deane FP, Marshall KL, Dalley A. Adolescents' suicidal thinking and reluctance to consult general medical practitioners. J Youth Adolesc. 2010 Apr;39(4):343-56. doi: 10.1007/s10964-009-9436-6. Epub 2009 Jul 15. PMID 20229227
- [Background] Norton AT, Herek GM. Heterosexuals' attitudes toward transgender people: findings from a national probability sample of US Adults. Sex Roles. 2013;68(11-12):738-753. doi:10.1007/s11199-011-0110-6
- [Derived] Martin A, Calhoun A, Paez J, Amsalem D. Destigmatizing perceptions about Black adolescent depression: randomized controlled trial of brief social contact-based video interventions. J Child Psychol Psychiatry. 2022 Nov;63(11):1270-1278. doi: 10.1111/jcpp.13570. Epub 2022 Jan 23. PMID 35066880